CLINICAL TRIAL: NCT06063824
Title: Feasibility and Acceptability of Single-Session Method of Levels Psychotherapy Within Primary Care
Brief Title: Feasibility & Acceptability of One-Session MOL Therapy in Primary Care
Acronym: FAOMTPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Finbar Dickinson, Chief Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 328697
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Other: Single-Session Method of Levels Intervention

INTERVENTIONS:
Other: Single-Session Method of Levels Intervention — This is a single session of method of levels psychotherapy delivered to patients of GP surgeries in primary care.

SUMMARY:
People sometimes wait a long time for psychological therapy and could have this sooner if they had only one session. This is because they may only require one session to meet their needs if this is provided quickly (Cannistrà et al., 2020) and may therefore require less therapy overall, and if they can access this, then services can run more efficiently, and overall capacity of services to offer therapy can increase.

Some therapies are hard to deliver in one session. But the method of levels (MOL) was conceived to be highly flexible with respect to session length and number of sessions, and this makes it easier to use in one-off sessions. It is designed to help people focus on problems they describe as being most relevant to them and to find their own solutions.

We want to know if we can give one session of MOL to people seeking help from their GP. We want to see if they find it helpful. So we need to find out if they want and attend the session and if they tell us about it.

This will help us decide whether to run a larger study exploring whether one session of MOL can help meet the goals of people seeking GP support. This could tell us whether MOL could help reduce waiting times.

We will ask people using GP surgeries if they want to participate. They will be offered one session of MOL with their usual support. We will ask them to complete questionnaires to see if they found the therapy helpful.

We will note how many participate, attend sessions, and complete questionnaires. We will check whether participants liked having MOL and will interview 10-12 of them to learn about what they thought.

The research will be funded by The University of Manchester.

DETAILED DESCRIPTION:
DESIGN This mixed-methods, randomised, controlled, single-arm acceptability and feasibility pilot trial study will use a within-subjects design featuring an experimental group (receiving one session of MOL alongside usual treatment) and no control group. The study will contain a qualitative element through the analysis of qualitative questionnaire and interview feedback.

The study's contingency plan involves adopting a case series methodology featuring a smaller number of participants (all of whom would be interviewed).

RECRUITMENT One group of participants will be recruited: service users of a GP surgery who will be offered one session of MOL. We intend to have 5 participating GP practices recruited for the study, and the plan is to recruit 25 patients. Of these, a further intention is to recruit 10 to 12 participants to attend an interview about their experiences of their session. The overall recruitment target is 25 participants across the 5 participating GP surgeries.

The contingency plan would involve recruiting a smaller number of participants, all of whom would be interviewed.

PROCEDURE Potential participants registered at a Manchester GP surgery will be asked if they would like to take part in the study. This will be through a verbal question from their GP, a letter sent to them by the practice manager, a poster, or a text from the GP surgery. Potential participants who express interest in taking part (by informing the surgery or their GP or by signing and submitting the consent to contact form on the website whose URL will be texted to them) will have an information sheet passed to them, and their contact details will be shared (by their GP if they express interest to their GP) with the trainee clinical psychologist.

After 24 hours have elapsed (to provide time to read the information sheet), these individuals will be contacted on a telephone used specifically for the study, whereupon the trainee clinical psychologist will check whether they still want to take part and will take consent if so. Consent will be taken by participants either signing an online consent form or by coming to the surgery to sign a physical consent form. At this point, the individual will complete an initial Core Outcome Measure and an initial screening tool (either in person if they have come to the surgery or over the phone if they have completed the consent form online). If participants score above 10 on the initial Core Outcome Measure, meet the inclusion criteria, do not meet the exclusion criteria, and express that they are having a difficulty with which they would like help, they will be recruited as a participant by the trainee clinical psychologist and told their participant ID number. At this point, a summary will be provided by their GP of any relevant risk information.

Participants will be asked to complete an initial set of outcome measures in addition to the completed Core Outcome Measure (i.e. a demographic questionnaire, the PHQ-9, the GAD-7 and the PSYCHLOPS), which they may complete and return on paper or electronically via Qualtrics (using their ID number), Qualtrics is an online survey system approved by the University of Manchester, and a unique link to the measures on Qualtrics will be emailed to each participant in order that they can complete these.

Participants will be given details of how to book an MOL session electronically. A random selection of 10-12 participants will be invited to attend post-session interviews, and more participants will be randomly selected and invited as needed until 10-12 participants have confirmed their willingness to attend interviews. The participants will be offered some potential appointment times (via email) from a list of those available, which will be allocated to whichever patients request a given slot first. The patients will then receive a confirmation of their appointment time via email.

At their appointment time, they will arrive at their GP surgery and will be collected from the waiting room by the trainee clinical psychologist. After an introduction, the single session of MOL will be carried out, which will be up to 60 minutes in length.

After their sessions have been completed, participants will be securely emailed a link to the qualitative questionnaire and the post-session quantitative measures. All participants will be contacted by the trainee clinical psychologist a week after their session, and during this conversation, the trainee clinical psychologist will check in with them, remind them that we are emailing them the link to the relevant questionnaires, and ask them to complete these.

At the post-session, semi-structured interview (which will take place at The University of Manchester, at the GP surgery at which the relevant participant is registered, or online via Microsoft Teams), a volunteer (who will have an honorary contract with The University of Manchester) will ask a series of questions to explore how the participants felt about their MOL session. These interviews will be transcribed by the trainee clinical psychologist.

Participants will be informed (by email) that they have not been selected for interview once the required number of participants have been successfully interviewed. The interviews will last up to 60 minutes approximately, and they will be recorded via Microsoft Teams if they take place virtually. Recordings will be deleted once their computer-generated transcripts (produced by Microsoft Teams) have been checked and used to enable complete transcription (and once the full transcripts have been checked and uploaded to the Research Data Storage Service). Computer-generated transcripts will be deleted once they have been checked.

The interviews will be conducted, recorded and uploaded to the Research Data Storage Service by the volunteer, and the interviews will take place after the MOL session has been taken place (and as soon as the participant and volunteer can find a mutually agreeable time).

For interviews taking place over Microsoft Teams, the plan is for video of the interviews to be recorded to ease the demands of transcription and to facilitate quicker uploading from the recording device to the Research Data Storage Service (and because Microsoft Teams cannot record audio without also recording video). If participants being interviewed via Teams do not wish to have video of the interview recorded, they may opt to turn their cameras off.

All participants will be invited to attend an interview in the event that the study's contingency plan is adopted.

ANALYSIS Data regarding the perceived acceptability of the single session of MOL will be obtained via the qualitative questionnaire that will be hosted on Qualtrics and by transcripts of participant interviews. All data collected will be pseudonymous. These data will be analysed thematically and in accordance with the principles detailed by Braun and Clarke (2019) - they will be perused carefully several times before codes are constructed and then arranged into possible themes. These will be continually reconsidered with reference to the qualitative data, and they will then be given names and definitions.

In order to convey information regarding feasibility, the percentages of participants who attend their session and who complete the questionnaires will be calculated and described, and means and standard deviations of questionnaire scores before and after the session of MOL will be presented. Figures concerning recruitment will also be described alongside these. If it is possible, we aim to estimate the effect size of single-session MOL in primary care by referring to the abovementioned means and standard deviations. A statistical analysis plan will be constructed and approved before data analysis begins.

In the event of the contingency plan being adopted, the revised research question would be "Does a single session of MOL delivered in primary care lead to a significant change in clinical outcome measures?" Therefore, statistical analysis would differ in these circumstances, and inferential statistics would be required.

ELIGIBILITY:
Inclusion Criteria:

Participants will:

1. Be able to speak and read English as a first language
2. Be registered at a participating GP surgery and be due to remain at the surgery until the study's completion
3. Provide informed consent to participate in the study
4. Be 18 years of age or older
5. Be able to complete outcome measures
6. Score above 10 on an initial core outcome measure
7. Express that they are having a difficulty with which they would like help.

Exclusion Criteria:

Participants will not:

1. Have a mental health difficulty with a confirmed and known organic or neurological foundation
2. Be under drug and alcohol services for a substance misuse problem
3. Be experiencing active psychosis
4. Be under secondary care services for a mental health difficulty
5. Express that they have had plans or intentions to end their life or to harm themselves over the month before recruitment
6. Express that they have attempted to harm themselves in the month before recruitment
7. Express that they have attempted to end their life in the year before recruitment
8. Be unable to travel to their GP surgery for their session.

Individuals who do not meet the study's inclusion criteria will be unable to participate in the research.

It is worth clarifying the reason that participants must be able to speak English as a first language. MOL involves the therapist asking their interlocutor to articulate their thoughts in the present moment. This could entail participants being interrupted in order that the therapist can ask about background thoughts that may be pertinent to the difficulty being discussed. The presence of English as a first language as an inclusion criterion is a way of ensuring sufficient English language skills for this process to take place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation-Outcome Measure | Up to 3 months

SECONDARY OUTCOMES:
Generalised Anxiety Disorder-7 | Up to 3 months
Patient Health Questionnaire-9 | Up to 3 months
Psychological Outcome Profiles | Up to 3 months
Demographic Questionnaire | Up to 3 months
Qualitative Questionnaire | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Wilbraham Surgery, Manchester, Greater Manchester
  - Cornishway Group Practice, Manchester, Greater Manchester

IPD SHARING:
Plan to Share IPD: No